CLINICAL TRIAL: NCT04536792
Title: A Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AG-946 in Healthy Volunteers and in Subjects With Sickle Cell Disease
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AG-946 in Healthy Volunteers and in Participants With Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG946-C-001; 2020-000691-38 (EudraCT Number)
Record Dates: First submitted 2020-07-15; First posted 2020-09-03 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers; Anemia, Sickle Cell
Keywords: Sickle Cell Disease; Healthy
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Single Ascending Dose (SAD) Phase (Experimental): Participants will receive a range of doses of AG-946 or placebo, orally, once on Day 1. AG-946 will be given under fasted or fed conditions.
  Interventions: Drug: AG-946; Drug: AG-946 Matched Placebo
- Part 2: Multiple Ascending Dose (MAD) Phase (Experimental): Participants will receive a range of doses of AG-946 or placebo, orally, once daily (QD) for 14 days or using an alternative dosing regimen for up to 28 days under fasted conditions.
  Interventions: Drug: AG-946; Drug: AG-946 Matched Placebo
- Part 3: Sickle Cell Disease (SCD) Phase (Experimental): Participants will receive a range of selected ascending doses of AG-946, orally, QD or using an alternative dosing regimen for 28 days.
  Interventions: Drug: AG-946

INTERVENTIONS:
Drug: AG-946 — AG-946, oral encapsulated coated-granules or tablets.
Drug: AG-946 Matched Placebo — AG-946 matched-placebo, oral encapsulated sugar spheres or tablets.
  Arms: Part 1: Single Ascending Dose (SAD) Phase; Part 2: Multiple Ascending Dose (MAD) Phase

SUMMARY:
The purpose of the study is to assess the safety and tolerability of AG-946 in healthy volunteers after oral administration of single ascending doses (SAD) and multiple ascending doses (MAD) of AG-946 over 14 or up to 28 days of dosing, and to identify a range of doses that are safe and pharmacologically active in participants with sickle cell disease. The SAD and MAD parts of the study will be randomized and double-blinded, and will assess the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of AG-946 as well as the effect of food (SAD only) on the pharmacokinetics (PK) of AG-946. The sickle cell disease (SCD) part of the study will be non-randomized and open-label, and is designed to identify 1 or more safe and tolerable dose(s) of AG-946 with potential activity in the treatment of participants with sickle cell disease (SCD).

ELIGIBILITY:
Inclusion Criteria:

SAD and MAD

* Participant is a healthy male or a female of nonchildbearing potential aged 18 to 55 years inclusive at the time of consent;
* Participant is able to understand and provide informed consent before the conduct of any protocol-specific screening procedures;
* Participant is willing and able to complete all study assessments and procedures;
* Participant has a bodyweight ≥50 kilograms (kg) and body mass index ≥18.5 and ≤32 kilograms per square meter (kg/m^2) at screening;
* Participant is in good general health with no clinically significant deviations from normal in screening medical history, physical examination, vital signs, or electrocardiogram (ECGs);
* Male participants must agree to be abstinent as part of their usual lifestyle or use contraception up to 90 days after last dose of study treatment;
* Participant is a non-smoker and has not used nicotine-containing products for at least 3 months prior to screening;
* Participant is willing to refrain from caffeine- or xanthene-containing products (eg, coffee, tea, cola, chocolate) for 48 hours before the first dose of study treatment through 7 days after the last dose of study treatment;
* Participant is willing to refrain from marijuana- or cannabinol-containing products for 7 days before admission through the final visit;
* Participant is willing to refrain from strenuous exercise starting 72 hours before admission through the final visit;
* Participant is willing to refrain from use of alcohol starting 7 days prior to admission through final visit;
* Participant agrees not to donate blood products for duration of study participation;
* Male participants must agree not to donate sperm for duration of study and for 90 days after the last dose.

Exclusion Criteria:

SAD and MAD

* Participant has previously enrolled in this study or has received an investigational drug with 3 months or 5 half-lives of the drug, whichever is longer, before the first dose of study treatment;
* Participant has previously received AG-946, except for participants who are dosing in the fed portion of the food-effect group;
* Participant has a heart rate-corrected QT interval (QTc) interval using Fridericia correction method (QTcF) >450 milliseconds (ms) at screening;
* Participant has used over-the-counter medication (excluding routine vitamins) within 7 days of the first dose of study treatment, unless agreed as not clinically relevant;
* Participant has used acetaminophen greater than 2 grams (g) in any 24-hour period up to 48 hours before the first dose of study treatment;
* Participants has clinically relevant screening laboratory tests results outside the normal range;
* Participant has a history of any relevant cardiovascular, renal, hepatic, chronic respiratory, or gastrointestinal disease; or hematologic, lymphatic, neurologic, endocrine, psychiatric, musculoskeletal, genitourinary, immunologic, dermatologic, or connective tissue disease or disorders;
* Participant has a history of serious mental illness, that includes, but is not limited to schizophrenia, bipolar disorder, or major depression;
* Participant has a history of any primary malignancy, except for basal cell or squamous cell carcinomas of the skin or cervical carcinoma in situ or other malignancies that have been curatively treated and with no evidence of disease for at least 5 years before screening;
* Participant has had surgery within 6 months before the first dose of study treatment;
* Participant has a preexisting condition that interferes with normal gastrointestinal anatomy or motility, and/or hepatic and/or renal function that could interfere with the absorption, metabolism, and/or excretion of the study treatment or has previously undergone cholecystectomy;
* Participant has systolic blood pressure (BP) ≥140 mm Hg or a diastolic BP of ≥90 mm Hg after 10 minutes rest at screening or before the first dosing of study treatment;
* Participant has medical or psychological condition deemed by the Investigator to be likely to interfere with the volunteer's ability to provide informed consent, cooperate, and/or participate in the study;
* Participant has a known allergy to any of the excipients or components of the study treatment;
* Participant tests positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody (Ab), or human immunodeficiency virus (HIV) infection -1 or -2 Ab;
* Participant has donated blood, had blood loss of more than 500 milliliters (mL), or has received transfusion of blood or plasma within 3 months before screening;
* Participant has a history of illicit drug abuse or alcoholism within the last 1 year before screening;
* Participant has consumed more than 21 units of alcohol a week within the last 1 year before screening;
* Participant has used prescription drugs within 2 weeks or 5 half-lives (whichever is longer) before the first dose of study treatment;
* Participant has a positive screen for drugs of abuse or urinary cotinine >200 nanograms per milliliter (ng/mL) at screening or admission; or a positive screen for alcohol (via urine analysis) at admission;
* Participant cannot communicate reliably with the Investigator;
* Participant cannot or is unlikely to cooperate with the requirements of the study;
* Participant has any conditions that, in the judgment of the Investigator, would make the volunteer unsuitable for enrollment or could interfere with the volunteer's participation in, or completion of, the study;
* Participant has known glucose-6-phosphate dehydrogenase (G6PD) deficiency or G6PD activity below the lower limit of the normal range at the screening visit.

Inclusion Criteria:

SCD

* Participant is a male or female aged 18 to 70 years inclusive at the time of consent;
* Participant has documented sickle cell anemia;
* Provided informed consent before the conduct of any protocol-specific screening procedures;
* If the participant is taking hydroxyurea (HU), L-glutamine, and/or crizanlizumab, the dose(s) must have been stable for at least 3 months before the first dose of AG-946;
* Participant must start or continue to take folic acid in the equivalent of at least 0.8 milligrams per day (mg/day) orally for the duration of the study, unless the Investigator considers dietary folic acid intake to be adequate;
* Participant has adequate organ function;
* Female participants who are of childbearing potential, must have negative pregnancy test during screening;
* Female participants who are of childbearing potential and male participants who have partners who are females of childbearing potential, must agree to be abstinent as part of their usual lifestyle or agree to use contraception from the time of providing informed consent to 28 days for women and 90 days for men after the last dose of AG-946;
* Participant must be willing to comply with all study procedures for the duration of the study.

Exclusion Criteria:

SCD

* Participant is a candidate for potentially curative treatment with bone marrow transplantation, and for whom participation in this study would delay or preclude such definitive treatment;
* Participant has documented history of pyruvate kinase deficiency (PKD) or red blood cell-specific form of pyruvate kinase (PKLR) mutation;
* Participant has had more than 6 vaso-occlusive crisis (VOCs) within the past 12 months that required a hospital, emergency room, or clinic visit;
* Participant is receiving regularly scheduled red blood cell (RBC) transfusion therapy, and/or has received a transfusion within the past 3 months before the first dose of AG-946;
* Participant is currently receiving treatment with voxelotor or any other agent intended to increase hemoglobin (Hb)-oxygen affinity;
* Participant has a significant medical condition that confers an unacceptable risk to participating in the study, and/or that could confound the interpretation of the study data as follows:

  1. Poorly controlled hypertension (defined as systolic BP >150 millimeters of mercury (mm Hg) or diastolic BP >90 mm Hg) refractory to medical management
  2. Any history of congestive heart failure; myocardial infarction; unstable angina pectoris; hemorrhagic, embolic, or thrombotic stroke; or recent venous thrombosis or pulmonary or arterial embolism
  3. Cardiac dysrhythmias judged as clinically significant by the Investigator
  4. QTcF >450 milliseconds (ms), unless related to right or left bundle branch block
  5. Clinically symptomatic cholelithiasis or cholecystitis
  6. History of drug-induced cholestatic hepatitis
  7. Iron overload sufficiently severe to result in a clinical diagnosis by the Investigator of cardiac, hepatic, or pancreatic dysfunction
  8. Have a diagnosis of any other congenital or acquired blood disorder, or any other hemolytic process as defined by a positive direct antiglobulin test, except for mild alloimmunization as a consequence of transfusion therapy
  9. Positive test for HBsAg, or positive test for HCV Ab with evidence of active virus infection
  10. Positive test for HIV-1 or -2 Ab
  11. Active infection requiring the use of parenteral antimicrobial agents or Grade ≥3 in severity
  12. Diabetes mellitus judged to be under poor control by the Investigator or requiring >2 antidiabetic agents, including insulin
  13. History of any primary malignancy, except for curatively treated nonmelanoma skin cancer, cervical or breast carcinoma in situ, prostate cancer, or other primary tumor treated with curative intent, no known active disease present, and no treatment administered during the last 3 years before Screening
  14. Unstable extramedullary hematopoiesis that could pose a risk of imminent neurologic compromise
  15. Current or recent history of a psychiatric disorder
* Participant is currently enrolled in another therapeutic clinical trial involving ongoing therapy with any investigational or marketed product or placebo;
* Participant has had exposure to any investigational drug within 3 months or 5 half-lives of the drug, whichever is longer, before the first dose of AG-946;
* Participant has had exposure to any investigational device or invasive procedure within 3 months before the first dose of AG-946;
* Participant has a history of major surgery within 6 months of providing informed consent;
* Participant has had a prior bone marrow or stem cell transplant;
* Participant is currently pregnant or breastfeeding;
* Participant has received medications that are strong inhibitors of permeability-glycoprotein (P-gp) within 5 days or a time frame equivalent to 5 half-lives (whichever is longer) before the first dose of AG-946;
* Participant has received hematopoietic stimulating agents within 28 days before the first dose of AG-946;
* Participant has a known allergy to any of the excipients found in AG-946.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
SAD and MAD: Number of Participants Who Experienced at Least One Adverse Event (AE), by Severity | SAD: Up to Day 13; MAD: Up to Day 49
SAD and MAD: Number of Participants Who Experienced at Least One AE Related to the Study Drug | SAD: Up to Day 13; MAD: Up to Day 49
SAD and MAD: Number of Participants Who Experienced at Least One Serious Adverse Event (SAE) | SAD: Up to Day 13; MAD: Up to Day 49
SAD and MAD: Number of Participants With Clinically Significant Laboratory Abnormalities, by Severity | SAD: Up to Day 13; MAD: Up to Day 49
SAD and MAD: Number of Participants With Clinically Significant Changes in Vital Signs and in Electrocardiogram (ECG) Parameters | SAD: Up to Day 13; MAD: Up to Day 49
SCD: Number of Participants Who Experienced at Least One AE, by Severity | Up to Day 56
SCD: Number of Participants Who Experienced at Least One AE Related to the Study Drug | Up to Day 56
SCD: Number of Participants Who Experienced at Least One SAE | Up to Day 56
SCD: Number of Participants With Clinically Significant Laboratory Abnormalities, by Severity | Up to Day 56
SCD: Number of Participants With Clinically Significant Changes in Vital Signs and in ECG Parameters | Up to Day 56

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) of AG-946 | SAD: Up to Day 8; MAD: Up to Day 49; SCD: Up to Day 56
  Cmax will be determined under fasted and fed conditions in SAD and under fasted conditions only in MAD and SCD.
Time to Reach Maximum Observed Concentration (Tmax) of AG-946 | SAD: Up to Day 8; MAD: Up to Day 49; SCD: Up to Day 56
  Tmax will be determined under fasted and fed conditions in SAD and under fasted conditions only in MAD and SCD.
Area Under the Plasma Concentration-Time Curve from Time Zero to Last Quantifiable Concentration (AUC0-t), Time Curve from Time Zero to Infinity (AUC0-∞), and Time Curve from Time Zero to Time tau Over the Dosing Interval (AUC0-τ) for AG-946 | SAD: Up to Day 8; MAD: Up to Day 49; SCD: Up to Day 56
  AUC0-t, AUC0-∞, and AUC0-τ will be determined under fasted and fed conditions in SAD and under fasted conditions only in MAD and SCD.
SAD: Apparent Clearance (CL/F) for AG-946 | SAD: Up to Day 8
  CL/F will be determined under fasted and fed conditions.
SAD: Apparent Volume of Distribution (Vd/F) for AG-946 | SAD: Up to Day 8
  V/F will be determined under fasted and fed conditions.
SAD: Total Amount of Drug Excreted in Urine from Time 0 to Time T (Aet) and from Time t1 to Time t2 (Aet1-t2) for AG-946 Under Fasted and Fed Conditions | Up to Day 3
SAD: Percentage Dose of Drug Excreted in Urine from Time 0 to Time t (fet) and from Time t1 to Time t2 (fet1-t2) for AG-946 Under Fasted and Fed Conditions | Up to Day 3
SAD: Renal Clearance (CLr) for AG-946 Under Fasted and Fed Conditions | Up to Day 3
Changes in the Concentration of 2,3-diphosphoglycerate (2,3-DPG) and Adenosine Triphosphate (ATP) in Whole Blood | SAD: Up to Day 13; MAD: Up to Day 49; SCD: Up to Day 56
Area Under the Effect Curve (AUEC) from Time zero to t for 2,3-DPG and ATP | SAD: Up to Day 13; MAD: Up to Day 49; SCD: Up to Day 56
SAD: Relative Bioavailability Comparing Fasted to Fed Conditions Determined from the PK Parameters of AG-946 | SAD: Up to Day 8
SCD: Change From Baseline in Hemoglobin (Hb) | Up to Day 56
SCD: Change From Baseline in Direct Bilirubin | Up to Day 56
SCD: Change From Baseline in Lactate Dehydrogenase (LDH) | Up to Day 56
SCD: Change From Baseline in Haptoglobin | Up to Day 56
SCD: Change From Baseline in Reticulocytes | Up to Day 56
SCD: Change From Baseline in Erythropoietin | Up to Day 56

CONTACTS AND LOCATIONS:
Locations (10):
- United States (8):
  - University of California San Diego, La Jolla, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - New York Presbyterian Hospital - Weill Cornell Medicine, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - PPD Development, LP, Austin, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center - USOR, Dallas, Texas
  - University of Texas Health Science Center of Houston, Houston, Texas
- Rigshospitalet, Department of Hematology, Copenhagen, Denmark
- Hospital Universitario Vall d'Hebron - PPDS, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No